CLINICAL TRIAL: NCT00589303
Title: Pacing and AV Node Ablation Compared to Drug Therapy in Symptomatic Elderly Patients With Atrial Fibrillation Clinical Trial (PACIFIC) - Pilot Study
Brief Title: AV Node Ablation and Pacemaker Therapy Compared to Drug Therapy for Atrial Fibrillation - Pilot Study
Acronym: PACIFIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Win K Shen MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-004554
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Atrial Fibrillation; Heart Failure; AV Node ablation; Cardiac pacemaker; Antiarrhythmic drug
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure | interventions — Metoprolol; Atenolol; Carvedilol; Verapamil; Diltiazem; Procainamide; Disopyramide; Propafenone; Sotalol; dofetilide; Amiodarone; Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Therapy (Active Comparator): FDA approved rate and rhythm control drugs
  Interventions: Drug: FDA approved rate and rhythm control drugs
- Atrioventricular Node (AVN) Ablation / Pacing (Active Comparator): AV Node ablation and device implant
  Interventions: Device: AV Node ablation and device implant

INTERVENTIONS:
Drug: FDA approved rate and rhythm control drugs — Any approved rate or rhythm control drugs for treatment of atrial fibrillation may be prescribed under the primary physician's discretion.
  Rate Control:
  Beta-Blocker:
  * metoprolol
  * atenolol
  * carvedilol
  Calcium Channel Blocker:
  * verapamil
  * diltiazem
  Rhythm Control:
  * procainamide
  * quinidine
  * disopyramide
  * propafenone
  * flecainide
  * sotalol
  * dofetilide
  * amiodarone
  Other Names: Lopressor; Toprol XL; Tenormin; Coreg; Isoptin; Verelan; Verelan PM; Calan; Bosoptin; Covera-HS; Cardizem; Pronestyl; Norpace; Rythmol; Betapace; Tikosyn; Cordarone; Pacerone
  Arms: Drug Therapy
Device: AV Node ablation and device implant — Pacing Systems:
  * Enpusle Premarket Approval Number (PMA#) P980035
  * EnRhythm PMA# P980035
  * Adapta PMA# P980035
  Cardiac Resynchronization Therapy (CRT) Pacing Systems:
  - InSync III/ Insync Maximo/InSyncII Marquis PMA# P010031
  Implantable Cardioverter-Defibrillator (ICD) Pacing Systems:
  * EnTrust PMA# P980016
  * Virtuoso PMA# P980016
  ICD CRT Pacing Systems:
  * InSync Maximo PMA# P980016
  * InSync Sentry PMA# P890003
  * Concerto PMA# P980016
  Arms: Atrioventricular Node (AVN) Ablation / Pacing

SUMMARY:
The purpose of this study is to determine whether early atrioventricular node (AVN) ablation with pacing device therapy will reduce death and hospitalization when compared to the conventional drug therapy in elderly patients with recurrent and symptomatic atrial fibrillation (AF).

DETAILED DESCRIPTION:
Epidemiologic studies have shown that 70-80% of patients with atrial fibrillation are older than 65 years of age. Drug therapy for atrial fibrillation is not effective or not tolerated in many elderly patients, for both rate or rhythm strategies. Preliminary data from AVN ablation and pacemaker therapy demonstrated this strategy is highly effective in controlling symptoms among patients who have failed numerous drug therapy. Quality of life is improved while hospital admission and office visits are reduced.

Pilot Study Design

* All patients will be 1:1 randomized to standard-care drug therapy (American College of Cardiology/American Heart Association Guideline, 2006) or AV node ablation and pacemaker therapy
* For patients randomized to AVN ablation, there will be a 1:1 sub-randomization to conventional right ventricular apex pacing or cardiac resynchronization therapy (biventricular pacing)
* All patients will be followed at 2 and 6 months from the time of randomization in the pilot study.
* A total of 60 patients from 5-15 clinical sites will be enrolled during an active recruiting period of 12 months for the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 65 years
* Paroxysmal, persistent, or permanent atrial fibrillation
* Index event of atrial fibrillation is documented on electrocardiogram or rhythm strip. Atrial fibrillation must be the qualifying event. Atrial flutter can have been present in the past, but it must not be considered the index arrhythmia.
* Paroxysmal atrial fibrillation episodes must be recurrent (two or more episodes in the past 6 months). At least one of the paroxysmal episodes must be "sustained", defined as lasting greater than 1 hour documented by a Holter monitor or by history in conjunction with an ECG or a rhythm strip.
* At least one attempt of unsuccessful drug therapy, either for rate, for rhythm, or for rate-and-rhythm control.
* Symptoms related to atrial fibrillation within the last 6 months
* Eligible for long-term treatment with both treatment strategies
* Must provide informed consent, Health Insurance Portability and Accountability Act (HIPAA) authorization, and be willing to comply with follow-up requirements.

Exclusion Criteria:

* Reversible causes of atrial fibrillation
* On heart transplant list
* Familial cardiac conditions with increased risk of sudden death
* Asymptomatic
* Medical condition limiting expected survival to be less than one year
* Contraindications to anticoagulation
* Pre-existing implanted pacemaker, implantable automatic cardioverter-defibrillator or cardiac resynchronization device.
* Pre-existing indication for permanent pacemaker, implantable automatic cardioverter-defibrillator or cardiac resynchronization device
* More than one attempt of drug therapy for rate, for rhythm, or for rate-and-rhythm control
* Planned major surgery within the next six months, including thoracic surgery
* Disability that would preclude collection of study data or have co-morbidity that would contraindicate device implantation
* Participated in another clinical trial within the previous 30 days using a therapeutic modality which could have potential residual effects that might confound the results of this pilot study
* Unable to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Win K Shen, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (5):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - The Heart Group, Evansville, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - Chattanooga Heart Institute, Chattanooga, Tennessee
- University of Calgary and Calgary Health Region, Calgary, Alberta, Canada

REFERENCES:
- [Background] Van Gelder IC, Hagens VE, Bosker HA, Kingma JH, Kamp O, Kingma T, Said SA, Darmanata JI, Timmermans AJ, Tijssen JG, Crijns HJ; Rate Control versus Electrical Cardioversion for Persistent Atrial Fibrillation Study Group. A comparison of rate control and rhythm control in patients with recurrent persistent atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1834-40. doi: 10.1056/NEJMoa021375. PMID 12466507
- [Background] Bradley DJ, Shen WK. Atrioventricular junction ablation combined with either right ventricular pacing or cardiac resynchronization therapy for atrial fibrillation: the need for large-scale randomized trials. Heart Rhythm. 2007 Feb;4(2):224-32. doi: 10.1016/j.hrthm.2006.10.016. Epub 2006 Oct 20. PMID 17275763
- [Background] Bradley DJ, Shen WK. Overview of management of atrial fibrillation in symptomatic elderly patients: pharmacologic therapy versus AV node ablation. Clin Pharmacol Ther. 2007 Feb;81(2):284-7. doi: 10.1038/sj.clpt.6100062. PMID 17259952
- [Background] Ozcan C, Jahangir A, Friedman PA, Patel PJ, Munger TM, Rea RF, Lloyd MA, Packer DL, Hodge DO, Gersh BJ, Hammill SC, Shen WK. Long-term survival after ablation of the atrioventricular node and implantation of a permanent pacemaker in patients with atrial fibrillation. N Engl J Med. 2001 Apr 5;344(14):1043-51. doi: 10.1056/NEJM200104053441403. PMID 11287974
- [Background] Gregoratos G, Abrams J, Epstein AE, Freedman RA, Hayes DL, Hlatky MA, Kerber RE, Naccarelli GV, Schoenfeld MH, Silka MJ, Winters SL, Gibbons RJ, Antman EM, Alpert JS, Gregoratos G, Hiratzka LF, Faxon DP, Jacobs AK, Fuster V, Smith SC Jr; American College of Cardiology/American Heart Association Task Force on Practice Guidelines/North American Society for Pacing and Electrophysiology Committee to Update the 1998 Pacemaker Guidelines. ACC/AHA/NASPE 2002 guideline update for implantation of cardiac pacemakers and antiarrhythmia devices: summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/NASPE Committee to Update the 1998 Pacemaker Guidelines). Circulation. 2002 Oct 15;106(16):2145-61. doi: 10.1161/01.cir.0000035996.46455.09. No abstract available. PMID 12379588
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for the Management of Patients with Atrial Fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Aug 15;114(7):e257-354. doi: 10.1161/CIRCULATIONAHA.106.177292. No abstract available. PMID 16908781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 sites: (Mayo Clinic in Scottsdale, Arizona; Mayo Clinic in Rochester, Minnesota; Oregon Health and Science University in Portland, Oregon; University of Calgary in Calgary, Alberta, Canada; and The Heart Group in Evansville, Indiana.
Groups:
- Atrioventricular Node (AVN) Ablation / Pacing: Atrioventricular Node ablation and device implant
Period: Overall Study
Arm/Group | Drug Therapy | Atrioventricular Node (AVN) Ablation / Pacing
Started | 14 | 13
Completed | 12 | 12
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Therapy | Atrioventricular Node (AVN) Ablation / Pacing | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 14 | 13 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
  Canada | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Hospitalization Within Six Months of Enrollment
Description: Number of patients who were hospitalized for cardiovascular problems within 6 months of enrollment.
Time Frame: Six months after enrollment
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Drug Therapy | Atrioventricular Node (AVN) Ablation / Pacing
Number analyzed (Participants) | 14 | 13
participants | 3 | 4

ADVERSE EVENTS:
Time Frame: All subjects had a follow up at 2 and 6 months.
Arm/Group | Drug Therapy | Atrioventricular Node (AVN) Ablation / Pacing
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 1/14 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Therapy (N=14) | Atrioventricular Node (AVN) Ablation / Pacing (N=13)
Fluid accumulation (General disorders) | 1 (2) | 1 (1)
Viral Pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Muscle Stimulation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Worsening Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Pneumothroax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lead Reposition (Cardiac disorders) | 0 (0) | 1 (1) — The lead to the pacemaker had to be repositioned.
Volume Depletion (Cardiac disorders) | 0 (0) | 1 (1) — Volume depletion is the loss of both water and salts from cell volume.
Dizziness (General disorders) | 0 (0) | 1 (1)
Left upper extremity swelling (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated when about half of the subjects were enrolled due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No